CLINICAL TRIAL: NCT00399594
Title: Investigating Non-response to Cardiac Resynchronization: Evaluation of Methods to Eliminate Non-response & Target Appropriate Lead Location (INCREMENTAL).
Brief Title: Effect of Targeting Left Ventricular Lead Position on the Rate of Response to Cardiac Resynchronization Therapy.
Acronym: INCREMENTAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Medtronic (Industry); Hoffmann-La Roche (Industry); Cambridge Heart Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Derek Exner, Professor and Canada Research Chair in Cardiovascular Clinical Trials, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAH 70-3402
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure, Congestive; Cardiac Pacing, Artificial; Defibrillators
Keywords: Mechanical dyssynchrony; Biventricular pacing; Cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Targeted LV lead placement
  Interventions: Procedure: A
- B (Active Comparator): Usual LV lead placement
  Interventions: Procedure: B

INTERVENTIONS:
Procedure: A — LV lead placement in region of latest mechanical velocity (tissue doppler)
  Arms: A
Procedure: B — LV lead placement in standard (lateral / posterolateral) position.
  Arms: B

SUMMARY:
Identifying & optimizing strategies to reduce the burden of heart failure is vital. Despite advances in pharmacotherapy, patients with heart failure are at high risk for death & hospitalization. Cardiac resynchronization therapy (CRT) synchronizes ventricular mechanical activity, improves cardiac output & reduces HF symptoms. However, ~50% of patients do not clearly respond to CRT. Sub-optimal placement of the LV pacing lead appears to be an important reason for non-response.

This study will assess whether targeted LV lead placement will result in an increased probability of CRT response at 52 weeks vs. usual (lateral wall) lead placement.

DETAILED DESCRIPTION:
Background. Identifying & optimizing strategies to reduce the burden of heart failure (HF) is vital. Despite advances in pharmacotherapy, patients with HF are at high risk for death & hospitalization. Over 25% of patients with systolic HF have dyssynchronous ventricular contraction that results in paradoxical septal motion, further impairing left ventricular (LV) function & HF progression. Cardiac resynchronization therapy (CRT) synchronizes ventricular mechanical activity, improves cardiac output & reduces HF symptoms. However, ~50% of patients do not clearly respond to CRT. Sub-optimal placement of the LV pacing lead appears to be an important reason for non-response.

Screening. Mechanical synchrony is vitally important in optimizing CRT response. Patients will be pre-screened with echocardiograms (echo) & CRT provided to only those with dyssynchrony. The predicted rate of CRT response in patients pre-screened for dyssynchrony is estimated at 65%.

CRT response. The combined use of a valid & simple measure of functional capacity with a reproducible measure of LV volume is optimal in identifying CRT responders. These outcomes will be assessed using the Specific Activity Scale & radionuclide angiography (RNA), respectively.

Primary hypothesis. Targeted LV lead placement will result in an increased probability of CRT response at 52 weeks vs. usual (lateral wall) lead placement. CRT response will be defined as ≥ 10% relative reduction in LV end systolic volume & ≥ 1 Specific Activity Scale class improvement.

ELIGIBILITY:
Inclusion Criteria:

* LV EF ≤ 0.40 measured within 3 months of enrollment,
* SAS class 3 or 4 symptoms indicative of moderate to severe functional capacity limitation due to heart failure within 1 month of enrollment.
* Confirmed dyssynchrony on screening echo (1.1.9), &
* On stable doses of ACE inhibitor or angiotensin II blocker & a beta-blocker for ≥ 2 months unless medically contra-indicated.
* Controlled heart rate if in permanent AF (resting <70 & maximal <120).

Exclusion Criteria:

* Unable or unwilling to provide informed consent,
* Medical condition other than heart failure likely to cause death < 1 year,
* Cardiac transplant planned within 6 months,
* Known contra-indication to transvenous CRT device implant (e.g., active sepsis, artificial tricuspid valve, known vascular occlusion that will prevent delivery of leads transvenously),
* Clinically significant myocardial infarction within last 2 months, or
* Coronary bypass graft surgery ≤ 2 months or coronary angioplasty ≤ 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in end systolic volume plus reduction in symptoms | over 12 months

SECONDARY OUTCOMES:
Minnesota Living with Heart Failure score. | Change over 12 months
Short form thirty six score. | Change over 12 months
Specific Activity Scale score. | Change over 12 months
New York Heart Association class. | Change over 12 months
Six minute walk distance. | Change over 12 months
LV volumes. | Change over 12 months
N-terminal pro-B-type natriuretic peptide. | Change over 12 months
Mortality | Study duration
Hospitalization | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: Derek V Exner, MD, MPH, Principal Investigator — Libin Cardiovascular Institute of Alberta, University of Calgary
Locations (3):
- Canada (3):
  - Foothills Hospital, Calgary, Alberta
  - London Health Sciences, London, Ontario
  - Quebec Heart Institute, Ste-Foy, Quebec